CLINICAL TRIAL: NCT03481231
Title: In Situ Immune Parameters and Their Prognostic Role on the Survival of Patients With Glioblastoma
Acronym: IMMUNOGLIO
Status: Completed | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00531-52
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma
Keywords: immunotherapy; tumors and blood samples
MeSH Terms: conditions — Glioblastoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — 24 ml blood sample + tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glioblastoma (GBM) is the most frequent brain tumor. Currently survival is poor and few treatments are available. Recent data show that there is no immune privilege of the central nervous system (CNS) and that GBM are invaded by effector CD8 T cells, letting us hypothesis that GBM growth is dependent of immunosurveillance.

The aim of this study is to better understand the antitumor immune response against GBM to unravel new effectors and immunosuppressive pathways important for the regulation of anticancer immunity and to discover new immune activating strategies with the objectives to isolate subgroups of GBMs that could benefit from an immunotherapy approach. To achieve this goal, GBM tumor samples and a blood sample will be collected during the initial tumor resection.

The sites involved in the recruitment of the patients will be the neurosurgical teams in Brussel, Dijon, Nantes and Padova.

DETAILED DESCRIPTION:
Primary objective :

The primary objective is to determine for each of the 3 molecular subtypes of glioblastoma the predictive performance on 1-year overall survival of in situ immune parameters

Secondary objectives :

To identify the best combination of in vivo immune parameters that is predictive of 1-year overall survival To determine the impact of immune parameters on overall survival Create a collection of biological samples

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed, brain tumor
2. Gross or near total resection of the contrast-enhancing tumor mass decides by the neurosurgeron.
3. Subjects ≥18 and ≤75 years of age at surgery
4. Patients must be able to understand and sign the informed consent documents indicating that they are aware of the investigational nature of this study.
5. Confirmation of the diagnosis of grade IV GBM by the local pathologist with an independent neuropathologist who will review this diagnosis
6. Primary therapy must consist of surgical resection with the intent for a gross or near total resection of the contrast-enhancing tumor mass, followed by conventional external beam radiation therapy and concurrent temozolomide chemotherapy.
7. Tumor biopsy for biological analysis has to be performed before using ultrasonic surgery

Exclusion Criteria:

1. Patient with other type of primary brain tumor or metastases
2. Patients with only biopsy performed for the diagnosis
3. Subjects under guardianship, curatorship or judicial protection
4. Female subjects who are pregnant or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a glioblastoma
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
overall survival | 24 months
  Determination for each of the 3 molecular subtypes of glioblastoma the predictive performance on 1-year overall survival of in situ immune parameters

CONTACTS AND LOCATIONS:
Locations (5):
- France (3):
  - Centre Georges François Leclerc, Dijon
  - CHU de DIJON, Dijon
  - CHU de Nantes, Saint-Herblain
- Italy (2):
  - Università di Florence, Florence
  - Azienda Ospedaliera Università di Padova, Padua